CLINICAL TRIAL: NCT03119480
Title: The Effect of Electronic Warning Systems in the Process of Diagnosis and Treatment of Patients With Acute Kidney Injury
Brief Title: Electronic Warning Systems in Diagnosis and Treatment of AKI
Status: Completed | Type: Observational
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Ding Feng, Kidney internal medicine professor, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Other Study IDs: AKI-2017-01
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Acute Kidney Injury
Keywords: Acute Kidney Injury; Electronic alerts
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hospital-acquired AKI: Adult patients with Hospital-acquired AKI
  Interventions: Device: electronic alerts

INTERVENTIONS:
Device: electronic alerts — electronic alerts for AKI

SUMMARY:
To set up electronic early warning system of AKI patients; To develop AKI's intervention, the follow-up process, and the renal physician is responsible for the implementation.

To Observe the method after implementing the treatment efficacy of AKI and the differences between the traditional treatment process.

DETAILED DESCRIPTION:
To set up electronic early warning system according to KDIGO AKI diagnosis standard, real-time monitoring of hospitalized patients with renal function data, real-time detection of AKI patients, notify the diagnosis of renal physician; To develop AKI's intervention, the follow-up process, and the renal physician is responsible for the implementation.

To Observe the method after implementing the treatment efficacy of AKI and the differences between the traditional treatment process.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants were adults aged 18 years or older who were in hospital with stage 1 or greater acute kidney injury as defined by Kidney Disease Improving Global Outcomes creatinine-based criteria.

Exclusion Criteria:

Exclusion criteria were initial hospital creatinine 4•0 mg/dL (to convert to μmol/L, multiply by 88•4) or greater, fewer than two creatinine values measured, inability to determine the covering provider, admission to hospice or the observation unit, previous randomisation, or end-stage renal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adult patients aged>18 years,with hospital-acquired acute kidney injury, from a university-affiliated hospital in Shanghai, China
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
all-cause mortality | at 7 days after alert
  death at 7 days after alert

SECONDARY OUTCOMES:
dialysis | at 7 days after alert
  dialysis at 7 days after alert
change in creatinine | at 7 days after alert
  relative maximum change in creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Feng Ding, PhD, Study Director — Division of Nephrology,Shanghai Ninth People's Hospital, School of Medicine, Shanghai Jiaotong University
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai, Shanghai Municipality, China